CLINICAL TRIAL: NCT03133819
Title: The Early Intervention and Prevention of Diabetes Foot
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CMRPG2F0171
Record Dates: First submitted 2017-01-10; First posted 2017-04-28 (Actual); Last update posted 2017-05-08 (Actual); Status verified 2016-05

CONDITIONS: Diabetes; Neuropathy, Polyneuropathy (Manifestation)
MeSH Terms: conditions — Diabetes Mellitus; Polyneuropathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Q-Sense_QST (TSA II) (Other): QST measurement will perform on the thenar eminence of the dominant hand and the lateral distal aspect of the foot dorsum of the same side.
  Using the method of limits, a threshold will determine as the average of four successive stimuli for cold and warmth sensation and two for heat pain.
  Interventions: Device: Q-Sense_QST (TSA II)

INTERVENTIONS:
Device: Q-Sense_QST (TSA II) — QST will perform using the Medoc device (TSA2001/VSA3001) following previous published procedures. The measurement will perform on the thenar eminence of the dominant hand and the lateral distal aspect of the foot dorsum of the same side.

SUMMARY:
Peripheral neuropathy is just assessed by determination of Vibration sensation, pressure sensation, superficial pain or temperature. The most commonly used technique for diagnosis of peripheral neuropathy is nervous conduction (NC) and electromyography (EMG). But EMG/NC is bothersome and techniques using electric currents to measure NC and needles to study muscle innervations are uncomfortable.

Quantitative NeuroSensory Testing (QST) is essential in the evaluation of small-caliber A-delta and C-fibers, the primary transmitters of thermal and pain sensation. QST can demonstrate neurosensory abnormalities when it is non-invasive test, selective to small fibers despite negative EMG/NCV finding.

The investigators predict QST can be used for the early diagnosis and follow-up of small-fiber neuropathy in diabetes patients. The investigators also predict the early evaluation of diabetes neuropathy with QST can reduce the diabetes patient progress to advance stage of DM foot or limb amputation.

DETAILED DESCRIPTION:
Patients will be divide into 4 groups (groups 1 to 4 will be divided by Q-Sense QST (TSA II) . The patient groups will be defined as the followings:

1. Group 1: 100 diabetes patients without neuropathy, Q-Sense normal.
2. Group 2: 100 diabetes patients with neuropathy, Q-Sense abnormal but no evidence of PAOD.
3. Group 3: 100 diabetes patients with neuropathy, Q-Sense abnormal , PAOD (＋), but no foot ulceration
4. Group 4: 100 diabetes patients with neuropathy, PAOD(＋) , and foot ulceration QST will perform using the Medoc device (TSA2001/VSA3001) following previous published procedures.

ELIGIBILITY:
Inclusion Criteria:

* Group 1: 100 diabetes patients without neuropathy, Q-Sense normal.
* Group 2: 100 diabetes patients with neuropathy, Q-Sense abnormal but no evidence of PAOD.
* Group 3: 100 diabetes patients with neuropathy, Q-Sense abnormal , PAOD (＋), without foot ulceration.
* Group 4: 100 diabetes patients with neuropathy, PAOD (＋), and foot ulceration.

Exclusion Criteria:

* Poorly controlled hypertension (SBP≥150 under regular medical treatment)
* Thyroid disease
* Pregnancy
* Have been diagnosed malignancy
* Liver cirrhosis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2016-11; Primary Completion 2019-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Glycohemoglobin (HbA1c) | month 0, 6, 12
  To see the correlation between diabetes neuropathy (by Q sense measurement) and glycemic control status ( at baseline, 6 months and 12 months).
Lipid profile | month 0,6,12
  To see the correlation between diabetes neuropathy (by Q sense measurement) and lipid profile ( at baseline, 6 months and 12 months).
Diabetes nephropathy ( macro-albuminuria (UACR ≧300 mg/g) ，micro-albuminuria (UACR: 30 - 300 mg/g)) | month 0,6,12
  To see the correlation between diabetes neuropathy (by Q sense measurement) and albuminuria status ( at baseline, 6 months and 12 months). Check the albuminuria status by the criteria (macro-albuminuria (UACR ≧300 mg/g) ，micro-albuminuria (UACR: 30 - 300 mg/g))
Peripheral arterial occlusive disease | month 0,6,12
  To see the correlation between diabetes neuropathy (by Q sense measurement) and severity of peripheral arterial occlusive disease ( at baseline, 6 months and 12 months).

SECONDARY OUTCOMES:
Diabetes foot | month 0, 6, 12
  To see the correlation between diabetes neuropathy (by Q sense measurement) and diabetes foot, foot ulceration ( at baseline, 6 months and 12 months).
major lower leg events ( lower leg amputation or revascularization) | month 0,6,12
  To see the correlation between diabetes neuropathy (by Q sense measurement) and major lower leg events including lower leg amputation or revascularization) ( at baseline, 6 months and 12 months).
Major cardiac events ( myocardial infarction, strokes and cardiac related death) | month 0,6,12
  To see the correlation between diabetes neuropathy (by Q sense measurement) and major cardiac events including myocardial infarction, strokes and cardiac related death)( at baseline, 6 months and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Kuei-Mei Chou, MD, Principal Investigator — Chang Gung Memorial Hospital, Keelung

IPD SHARING:
Plan to Share IPD: No